CLINICAL TRIAL: NCT02323802
Title: Diet Therapy Versus Prescriptive Educational Group Intervention in Overweight / Obese Patients at First Episode of AMI: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Chiara Muggia, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMI-Obesity
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Obesity /Overweight; Acute Myocardial Infarction (STEMI/ NSTEMI)

ARMS (2):
- educational group intervention (Experimental): The group educational food intervention: it provides the delivery of information leaflet and inclusion in groups on a weekly basis for the first 3 meetings, and then, there are other 2 meetings on the third and sixth month by the AMI.
  The meetings will cover education to self-nutrition, physical activity and learning techniques for stimulus control and management of high-risk situations.
  Interventions: Behavioral: educational group intervention
- prescriptive diet (Active Comparator): An objectives food scheme elaborated for each patients will provide the reduction in caloric intake (equivalent to 500-600 calories in deficit if compared to the estimated daily requirement, based on the RDAs) and a reduced intake of lipids, which does not exceed 30% of total calories introduced, with a contribution of saturated fat no more than 7-9% .
  Interventions: Behavioral: prescriptive diet

INTERVENTIONS:
Behavioral: educational group intervention
  Arms: educational group intervention
Behavioral: prescriptive diet
  Arms: prescriptive diet

SUMMARY:
Results after interventions on lifestyle in the secondary prevention of ischemic heart disease are not always consistent, and the Guidelines multidisciplinary measures aren't easily achievable.

Therefore, the purpose of this research project is the identification of an interventional approach to effective secondary prevention and realistic feasibility, in a field of multifactorial risk. The study is open to patients who totaled a double chronic disease, obesity/overweight and coronary heart disease, and who experienced a first event of ischemic cardiac infarction (AMI). The aim is to evaluate the effectiveness of a group educational intervention in a sample of overweight and obese patients (BMI > 24.9) incurred in a first episode of acute myocardial infarction (non-STEMI and STEMI), comparing with the classic approach of prescriptive diet therapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects of both sexes and age ≥ of 18 years consecutively admitted to the Coronary Unit of IRCCS Foundation Policlinico S. Matteo, at first episode of STEMI or non-STEMI AMI, with BMI greater than 24.9.

Exclusion Criteria:

Patients who can not provide informed consent (because illiterate or with significant language barrier or severe deficit/cognitive decays). Subjects with diseases and/or disabling organ damage. Subjects affected by active neoplasm. Individuals who have submitted arhythmic complications in acute and/or heart failure, or people referring to post-AMI residential rehabilitation. Subjects that are carriers of severe psychiatric disorders diagnosed by DSM-V -TR.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
reduction of body weight | 6 months
  The proportion of subjects with a 10% reduction in body weight at 6 months

SECONDARY OUTCOMES:
Reduction of reinfarction and revascularization | 1 year
general and specific mortality | 1 year
  relative risk of death from all causes and from ischemic heart disease (no. of overall deaths and cardiovascular causes).
quality of life | 6 months
  quality of life (assessed by SF-36 questionnaire at baseline and 6 months after infarction).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Internal Medicine Department, Clinica Medica II, IRCCS San Matteo Foundation, Pavia, PV
  - Cardiology department, Pavia